CLINICAL TRIAL: NCT02949531
Title: Randomised, Cross Over, Single Blind, Control Trial of Short Term Oxygen Use During Cycle Ergometry in Patients With Chronic Heart Failure With Preserved Ejection Fraction
Brief Title: Use of Oxygen in Heart Failure With Preserved Ejection Fraction
Acronym: STOP-EF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R1965
Record Dates: First submitted 2016-10-03; First posted 2016-10-31 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2016-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 21% oxygen (Active Comparator): room air will be delivered via Venturi mask during cycle ergometry
  Interventions: Drug: oxygen
- 28% oxygen (Active Comparator): 28% oxygen will be delivered via Venturi mask during cycle ergometry
  Interventions: Drug: oxygen
- 40% oxygen (Active Comparator): 40% oxygen will be delivered via Venturi mask during cycle ergometry
  Interventions: Drug: oxygen

INTERVENTIONS:
Drug: oxygen

SUMMARY:
Oxygen is routinely given to patients with common conditions such as COPD and heart failure. There is no evidence behind giving oxygen to patients specifically in heart failure due to a stiff heart.

This study aims to explore the effect oxygen has on the ability of patients with chronic heart failure and the ability to exercise. Other common variables will be assessed such as heart rate and blood pressure to observe the response to varying concentrations of oxygen.

The concentrations chosen are commonly offered in hospitals and indeed are being delivered through standard equipment found in all hospitals in the country.

It is hoped that studying the effect of short term oxygen on patients with heart failure will help to identify the effectiveness of oxygen in longer term therapy for patients who are often breathless with a decreased exercise tolerance.

DETAILED DESCRIPTION:
Many patients with reduced exercise tolerance have a preserved left ventricular function. These patients are labelled as having heart failure with preserved ejection fraction (HeFPEF), when the combined use of echocardiography and biochemistry. The prevalence and the incidence of HeFPEF are on the increase and currently it accounts for around 50% of all patients diagnosed with HF. The last twenty years of research has led to great improvement in available treatments for heart failure with reduced ejection fraction (HeFREF); however, current guidelines only suggest diuretics to improve symptoms of those patients with HeFPEF: clinical trials of several pharmacological interventions have failed to show convincing reductions in morbidity or mortality for patients with HeFPEF.

The effect of oxygen therapy on exercise capacity has remained poorly understood in HeFREF and, at the time of writing this study, it has never been explored in HeFPEF. The investigators recently completed a study showing an increase in exercise time, exercise load at peak exercise and peak metabolic equivalent on cycle ergometry with 28% oxygen supplementation and further increments when 40% oxygen supplementation was used in patients with heart failure with reduced ejection fraction.

The investigators aim to improve exercise time in patients with HeFPEF with oxygen supplementation. Identifying the correct dose of oxygen will be a further aim to avoid hyperoxygenation but provide adequate oxygen to improve exercise tolerance.

Patients will be identified from heart failure clinics and will be invited for screening visit. Eligible patients will have three treatment visit at least one week apart (each visit with a different oxygen concentration i.e room air, 28% and 40% oxygen, randomly determined by sealed envelopes)

Patients will use standard cycle ergometry to exercise and work load will be increased every minute by 5-10 watts. Patients will be encouraged to cycle until tired. At the end of cycling, exercise time, peak metabolic equivalent, work load, shortness of breath score will be noted at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Over 50 years of age and able and willing to give consent
* Have signs and/or symptoms of heart failure
* Left ventricular ejection fraction > 45%
* NT-pro BNP > 220 pg/ml (in the previous 12 months)
* On any diuretic

Exclusion Criteria:

* Unable or unwilling to give consent
* Recent (<1 month) acute myocardial infarct or cerebrovascular event
* Significant renal dysfunction (eGFR <30 ml.min-1.1.73m-2)
* Significant anaemia (Haemoglobin < 100 g.L-1)
* Systolic blood pressure <90 mmHg, or >180 mmHg
* Severe mitral or aortic valve disease
* Diagnosis of severe chronic lung disease
* Involvement in another medicinal trial within the past four weeks
* Unable to use cycle
* Any planned admission in the following 3-4 weeks (patient can be reconsidered for enrolment after planned admission)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
change in exercise time with the use of 21%, 28% and 40% oxygen | at 3 weeks
  the total time cycled in each arm

SECONDARY OUTCOMES:
change in shortness of breath with the use of 21%, 28% and 40% oxygen | at 3 weeks
  shortness of breath measured using BORG score
change in Peak metabolic equivalent with the use of 21%, 28% and 40% oxygen | at 3 weeks
  measured using standard peak metabolic equivalent

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Clark, Principal Investigator — Castle Hill Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah P, Pellicori P, Rimmer S, Rigby AS, Clark AL. Effect of increased inspired oxygen on exercise performance in patients with heart failure and normal ejection fraction. Int J Cardiol. 2018 Oct 1;268:166-169. doi: 10.1016/j.ijcard.2018.05.029. Epub 2018 May 24. PMID 29803343